CLINICAL TRIAL: NCT04639557
Title: Building Regulation in Dual Generations - A Telehealth Parenting Program for Depressed Mothers of Preschoolers, Matched With Dialectical Behavior Therapy Skills
Brief Title: Building Regulation in Dual Generations - Telehealth Model
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Research Manitoba (Other); Centre for Addiction and Mental Health (Other); University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRIDGEV2.0
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2020-11

CONDITIONS: Maternal Depression; Child Development; Child Mental Health

STUDY DESIGN:
Intervention Model Description: The study will recruit a group of mother-child dyads in which the mother meets the current criteria for major depressive disorder. Mothers will be randomly assigned to one of two intervention arms, which will occur concurrently over 16-weeks. Both arms incorporate intervention materials from Dialectical Behavior Therapy (DBT) and parent skills training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Intervention (Experimental): Mothers in this group will participate in 16, once per week, scheduled 2-hour virtual group therapy sessions through Zoom for Healthcare. These sessions will include both visual media (e.g., presentations, recorded examples of skills), and discussions. A technician will be present in the virtual group therapy session to manage the technical component. These sessions will be supplemented with a 1-hour drop-in session moderated by a facilitator each week in which participants will be able to clarify topics for that week, discuss the material in more depth, and/or connect with other participants to share about the skill practice.
  Interventions: Behavioral: BRIDGE Therapy Program
- Therapy Intervention Pre-recorded (Experimental): Mothers in this group will have access to short pre-recorded videos of the presentations with facilitator commentary (i.e., 10-12 minutes) with additional video material as warranted each week (e.g., recorded examples of skill practice) for a maximum of 30-minutes of material per week. This arm will also have a 1-hour drop-in session each week with a group facilitator to moderate homework check-ins and discussion of the material.
  Interventions: Behavioral: BRIDGE Therapy Program

INTERVENTIONS:
Behavioral: BRIDGE Therapy Program — The BRIDGE Therapy Program is a novel manualized therapy that incorporates key parenting concepts and related Dialectical Behavior Therapy (DBT) modules. The primary aim of the program is to promote self-regulation in the mother-child dyads. There are two components of the program: 1) the DBT section, which will follow the DBT Skills Training Manual 2nd Edition and target maternal mental health symptomology, and 2) the parent skill training materials, which have been designed to correspond to the four core DBT modules (i.e., Mindfulness, Emotion Regulation, Distress Tolerance, and Interpersonal Effectiveness) and to promote self-regulatory skill development and a positive parent-child relationship.

SUMMARY:
Families who experience maternal mental illness and a variety of chronic stressors are currently underserved by the parenting programs. The investigators propose that impairments in maternal self-regulation, which result in unsupportive parenting, directly impact children's own self-regulation and neurobiology, leading to risk for intergenerational transmission of mental illness. The objective of this study is to develop and evaluate a program that is targeted at improving underlying self-regulatory mechanisms in both mothers with depression and their 3- to 5-year-old children. It is hypothesized that children exposed to maternal mental illness will have greater self-regulatory deficits across emotional and behavioural domains compared to children not exposed to mental illness. The effects of maternal mental illness are expected to be compounded for children of mothers reporting a higher degree of chronic stressors, including poverty, housing instability, violence, and low social support. Further, it is hypothesized that taking a dual-generation intervention approach to addressing self-regulatory mechanisms underlying psychopathology at the level of the mother, child, and dyad (i.e. parenting interactions) will improve both maternal capacities and child outcomes. A feasibility study has been conducted in-person (NCT04347707). Results from this trial showed positive effects on child and mother well-being as well as parenting skills. Our current study will be conducted remotely due to the COVID-19 pandemic to adhere to public health guidelines to reduce in-person contact and physical distance. The objectives for this study are two-fold: 1) establish a better understanding of the self-regulatory processes that are altered in preschool-aged children exposed to maternal mental illness, and determine the mediating role of parenting behaviours, as well as the moderating impact of chronic stress exposure; and 2) evaluate a novel dual-generation intervention for mothers with mental illness using a virtual format and their 3- to 5-year-old children based on existing gold-standard evidence-based approaches.

ELIGIBILITY:
Inclusion Criteria:

* Must have a 3-5 year old child
* The child must not have a diagnosed developmental delay
* Must have full or joint custody of the child
* Must meet current criteria for a Major Depressive Episode
* Must be 18 years of age

Exclusion Criteria:

* Child is outside of the 3-5 year old age range
* The child has a diagnosed developmental delay
* Mother does not have full or joint custody of the child
* Mother did not meet current criteria for a Major Depressive Episode (control group)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only mothers are eligible to participate.
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Maternal Depression from pre-intervention to post-intervention - Beck Depression Inventory | The Beck Depression Inventory will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time once again after the program is complete (approx. 20 weeks after Time 1).
  21-item self-report inventory to measure symptoms and characteristics of depression. Participants respond to statements on a 0-3 Likert scale. Higher scores indicate higher depression symptoms. The highest possible score is 60 and lowest possible score is 0.
Change in Maternal Emotion Regulation pre-intervention to post-intervention - Difficulties in Emotion Regulation Scale | The Difficulties in Emotion Regulation Scale will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  18-item self-report questionnaire with 6 sub-categories to measure emotion regulation. Participants respond to items on a 5-point Likert scale. Higher scores suggest more severe problems with emotion regulation. The highest possible score is 90 and the lowest possible score is 18.
3. Change in Parenting Stress from pre-intervention to post-intervention - Parenting Stress Index (Short form) | The Parenting Stress Index (short form) will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  36-item self-report measure filled out by parents to measure stress level within the context of parenting. Participants respond to items on a 5-point Likert scale. There are 3 sub categories. Responses to each item in a sub-category are totalled and then the 3 subcategory scores are summed to represent a total stress score. Higher scores indicated higher levels of parenting stress. Normal scores fall within the 15th to 85th percentile, and scores above the 85th percentile represent clinically elevated levels of stress.

SECONDARY OUTCOMES:
Change in the Child Behaviour Checklist from pre-intervention to post-intervention | The Child Behaviour Checklist will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  103-item questionnaire that asks parents to describe their child's behavioural and emotional problems within the past 2 months.
Change in Parental Sensitivity from pre-intervention to post-intervention | Parent-child interactions will be observed and video coded at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  Parent-child interactions will be video recorded after the child has participated in an acute stressor task. The interaction will be coded to measure levels of parental sensitivity using a novel coding scale (no established range).

OTHER OUTCOMES:
Change in Child Cognitive Function from pre-intervention to post-intervention - Exploratory Outcome | Child cognitive function will be assessed at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  Child cognitive function will be assessed with behavioural regulation tasks. Specifically, children will participate in the child version of the Stroop task, in which they will be required to say the opposite in response to pictures of Day/Night images and Happy/Sad faces.
2. Change in Child Stress System Reactivity and Recovery from pre-intervention to post-intervention - Exploratory Outcome | Child stress system reactivity and recovery will be measured at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  Child stress system reactivity will be measured through heartrate and salivary cortisol. Children will participate in an acute stressor task during which they will be wearing a FitBit heart rate monitor that will be recording their heartrate during the task. Salivary cortisol will also be collected immediately before the acute stressor, immediately after, and then 15, 30, and 45 minutes after.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manitoba - Department of Psychology, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Paton A, Stienwandt S, Penner-Goeke L, Giuliano RJ, Roos LE. Feasibility of an Online Acute Stressor in Preschool Children of Mothers with Depression. Dev Psychobiol. 2024 Sep;66(6):e22520. doi: 10.1002/dev.22520. PMID 38923527